CLINICAL TRIAL: NCT02087436
Title: Taperloc Complete Microplasty vs Taperloc Complete Standard: Randomized Controlled Study on Bone Mineral Density
Acronym: taperloc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INT.CR.GH3.13
Record Dates: First submitted 2014-01-14; First posted 2014-03-14 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2019-07

CONDITIONS: Osteoarthritis; Avascular Necrosis; Traumatic Arthritis; Rheumatoid Arthritis; Legg-Perthes Disease
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid; Legg-Calve-Perthes Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taperloc Complete Standard (Active Comparator): Group one will receive a total hip replacement with Taperloc Complete Standard. Taperloc Complete Standard is designed after the philosophy of a flat tapered wedge. It has evolved to incorporate the Reduced Distal and Microplasty stems to better address all patient anatomies, and facilitate multiple surgical techniques.
  Interventions: Device: Taperloc Complete Standard
- Taperloc Complete Microplasty (Active Comparator): Group one will receive a total hip replacement with Taperloc Complete Microplasty.Taperloc Complete Microplsty cementless stem is designed to transmit load to the proximal femur, thereby preserving bone density, and preventing long term instability and loosening secondary to proximal bone resorption.
  Interventions: Device: Taperloc Complete Microplasty

INTERVENTIONS:
Device: Taperloc Complete Microplasty — Taperloc Complete Microplsty cementless stem is designed to transmit load to the proximal femur, thereby preserving bone density, and preventing long term instability and loosening secondary to proximal bone resorption.
  Arms: Taperloc Complete Microplasty
Device: Taperloc Complete Standard — Taperloc Complete Standard is designed after the philosophy of a flat tapered wedge. It has evolved to incorporate the Reduced Distal and Microplasty stems to better address all patient anatomies, and facilitate multiple surgical techniques.
  Arms: Taperloc Complete Standard

SUMMARY:
The primary purpose of this study is to measure the postoperative changes in bone mineral density, comparing the Taperloc Complete Reduced Distal Microplasty stem and the standard length Taperloc Complete Reduced Distal stem.

DETAILED DESCRIPTION:
The Taperloc Microplasty cementless stem is designed to transmit load to the proximal femur, thereby preserving bone density, and preventing long term instability and loosening secondary to proximal bone resorption. The primary aim of this study is therefore to compare the postoperative changes in bone density with the Taperloc Microplasty stem, using the standard length Taperloc stem as a control.

In addition, the Taperloc stem has historically had a neck angle of 138°. There have been criticisms that this neck angle is too high for the typical Korean population. The newer Taperloc Complete system (both Microplasty and standard length) has a neck angle of 133°. A secondary aim is Occurrence ratio of thigh pain difference between Microplasty and standard stem in Korean Population

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for primary Total Hip Replacement

Patients with degenerative joint disease (inflammatory or non-inflammatory) or any of the composite diagnoses of:

1. Osteoarthritis
2. Avascular necrosis
3. Legg Perthes
4. Rheumatoid Arthritis
5. Diastrophic variant
6. Fused hip
7. Sequelae of Slipped capital epiphysis
8. Traumatic arthritis
9. Patients aged over 20
10. Patients must be able to understand instructions and be willing to return for follow-up

Exclusion Criteria:

* Absolute contraindications include: infection, sepsis, and osteomyelitis.

Relative contraindications include:

1. uncooperative patient or patient with neurologic disorders who are incapable of following directions,
2. Small Femoral canal

2) Severe osteoporosis (Patients over 65 years old) 3) metabolic disorders which may impair bone formation, 4) osteomalacia, 5) distant foci of infections which may spread to the implant site, 6) rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram, and 7) vascular insufficiency, muscular atrophy, or neuromuscular disease. 8) pregnancy 9) Fracture of the pelvis 10) Subcapital fractures

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | 1 year
  evaluate bone mineral density around the implant

SECONDARY OUTCOMES:
Radiographic Evaluation, | 2 years
  Radiographic measurements of stability and fixation
VAS Score | 2 years
  The measurement of pain intensity
Modified Harris Hip Score | 2 years
  * Over all Survivorship
  * Harris Hip Score
Radiographic Evaluation | 1 year
  Radiographic measurements of stability and fixation
Radiographic Evaluation | 6 Weeks
  Radiographic measurements of stability and fixation
VAS Score | 1 year
  The measurement of pain intensity
VAS Score | 6 Weeks
  The measurement of pain intensity
VAS Score | 6 Months
  The measurement of pain intensity
Modified Harris Hip Score | 1 year
  * Over all Survivorship
  * Harris Hip Score
Modified Harris Hip Score | 6 Months
  * Over all Survivorship
  * Harris Hip Score
Bone Mineral Density | Immediate post-op(2 - 4Weeks)
  * Two X-ray beams with different energy levels are aimed at the patient's bones.
  * DEXA
  * evaluate the bone mineral density around the implant

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Chan Ha, PHD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Young-Kyun Lee, PHD, Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Chung-Ang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT02087436/Prot_SAP_000.pdf